CLINICAL TRIAL: NCT00102830
Title: A Phase 1 Study Evaluating the Safety, Pharmacokinetics and Pharmacodynamics of AMG 386 in Adult Patients With Advanced Solid Tumors
Brief Title: Study Evaluating AMG 386 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Purpose: Treatment
Other Study IDs: 20040169
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Tumors
Keywords: Solid Tumor; Metastatic Cancer; Advanced Solid Tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — trebananib

INTERVENTIONS:
Drug: AMG 386

SUMMARY:
The purpose of this study is to test the safety, tolerability and pharmacokinetic (PK) profile of AMG 386 after intravenous administration in adult subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria: - Have evaluable disease - Must be able to undergo MRI evaluation:

1. Must not have cardiac pacemakers or neurostimulators not specifically approved for use in the MRI environment;
2. Must not have metal implants, other than those approved as safe for use in MRI;
3. Must not be claustrophobic or have physical characteristics that will preclude undergoing MRI; - Subjects enrolling to the Dose Expansion Cohort must have at least one tumor that is amenable to DCE-MRI evaluation (e.g., greater than or equal to 3 cm lesion outside the thoracic cavity) - Have Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2 - Adequate hematologic, renal and hepatic function Exclusion Criteria: - Presence of untreated CNS metastasis or symptoms of brain metastases - Presence of leukemia or myelodysplastic syndrome - History of high-dose chemotherapy requiring bone marrow or peripheral stem cell support - Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure [NYHA greater than class II], uncontrolled hypertension [diastolic greater than 85 mmHg; systolic greater than 145 mmHg] or cardiac arrhythmia) - History of arterial thrombosis (i.e., stroke, transient ischemic attack or myocardial infarction) within 6 months of study day 1 - History of bleeding diathesis or hypercoagulopathy within 6 months of study day 1 - Active peptic ulcer disease or gastritis - Unresolved toxicities from prior anti-cancer therapy, excluding alopecia - Anti-tumor treatment within 3 weeks of study day 1. If anti-tumor treatment was an antibody therapy, the interval must be 6 weeks - Anticoagulation therapy, except a low dose of Coumadin™ (less than 2 mg) for prophylaxis against central catheter-related thrombosis - Major surgery within 4 weeks of study day 1 - History of allergic reaction to bacterially produced proteins - Known positive test for human immunodeficiency virus (HIV) infection, hepatitis C virus or chronic hepatitis B infection - Pregnant or breastfeeding - Not using adequate contraceptive precautions, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Adverse events, clinically significant changes in laboratory results, ECG, and vital signs, to be measured throughout the study.
Pharmacokinetic Profile of AMG 386 - blood levels of AMG 386 to be measured throughout the study.

SECONDARY OUTCOMES:
Changes in DCE-MRI imaging results measured at baseline, Week 1, and Week 4.
Changes in blood levels of angiogenic cytokines measured at baseline, Day 3, Weeks 2, 4, 10, and every 8 weeks thereafter.
Anti-AMG 386 antibody formation measured at baseline, weeks 2, 4, 6, and every 4 weeks thereafter.
Tumor response measure by CT scan at baseline, Week 4, and every 8 weeks thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Lu JF, Rasmussen E, Karlan BY, Vergote IB, Navale L, Kuchimanchi M, Melara R, Stepan DE, Weinreich DM, Sun YN. Exposure-response relationship of AMG 386 in combination with weekly paclitaxel in recurrent ovarian cancer and its implication for dose selection. Cancer Chemother Pharmacol. 2012 May;69(5):1135-44. doi: 10.1007/s00280-011-1787-5. Epub 2012 Jan 1. PMID 22210018
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_65_AMG_386_20040169.pdf